CLINICAL TRIAL: NCT06727006
Title: Stroke, Thrombolysis and Rescue Stenting
Brief Title: Rescue Stenting and Intravenous Thrombolysis in Patients with Large Vessel Ischemic Stroke
Acronym: STARS
Status: Recruiting | Type: Observational
Sponsor: ASST Santi Paolo e Carlo (Other)
Responsible Party: Principal Investigator, Elena Ballabio, Full time dependent Neurologist Doctor. Working at neurologica department at ASST-Santi Paolo e Carlo at Milan-Italy, ASST Santi Paolo e Carlo
Other Study IDs: STARS12042023
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Large Vessel Occlusion; Stroke Acute; Thrombolysis; Rescue Stenting
Keywords: Rescue stenting; Thrombolysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute large vessel occlusion stroke undergoing rescue stenting

SUMMARY:
Intravenous thrombolysis (IVT) and mechanical thrombectomy (MT) are the standard of care for treating selected patients with acute large-vessel occlusion stroke (LVOS). Successful revascularization is strongly correlated with favorable outcomes. Nevertheless, recanalization failure with stent retrieval and contact aspiration has been observed in up to 29% of patients. If primary thrombectomy fails to achieve recanalization, rescue stenting (RS) has proven to be a feasible rescue therapy. Currently, approved evidence-based alternatives for LVOS patients who have failed MT are lacking, but permanent stenting is suggested as a rescue treatment in expert consensus statements.

Dual antiplatelet therapy (DAPT), typically consisting of clopidogrel and aspirin, is recommended after stent implantation to reduce the risk of stent thrombosis; however, these medications are not suitable in the acute setting, and optimal platelet inhibition strategies remain unclear. Glycoprotein (GP) IIb/IIIa receptor inhibitors have intravenous administration, a rapid onset of action, and their effects subside within a few hours after discontinuation. For these reasons, an increasing number of studies have investigated their use in conjunction with primary stenting for acute stroke. Currently, there is no evidence supporting the superiority of any particular antithrombotic strategy, so decisions are guided by clinical judgment.

An additional challenge for clinicians arises when IVT is combined with stenting. Stroke guidelines recommend starting antiplatelets 24 hours after IVT and the risk associated with antithrombotic therapy within the first 24 hours after IVT remains uncertain.

This is multicenter, prospective, observational study of patients with LVOS undergoing mechanical thrombectomy and rescue stenting. The aim of this study is to evaluate real-world antithrombotic strategies in emergency stenting, particularly in patients treated with IVT, and to assess the safety of emergent stenting following intravenous thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with large vessel occlusion strokes undergoing thrombectomy and rescue stenting within 24 hours of stroke onset
* Patients ≥ 18 years of age

Exclusion Criteria:

* Patients < 18 years
* Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with acute large vessel occlusion strokes undergoing rescue stenting in participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of symptomatic cerebral hemorrhage | 24 hours
  Symptomatic intracerebral hemorrhage (sICH) was defined as a worsening in National Institutes of Health Stroke Scale (NIHSS) score of ≥4 points within 24 hours with evidence of any hemorrhage on follow-up neuroimaging.

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) | 3 months
  mRS, a 6-level, clinician-reported, measure of global disability, with 0 being no symptoms and 6 being death. mRS is dichotomized where good functional outcome is a score 0 - 2 and poor functional outcome 3-6.

OTHER OUTCOMES:
Rate of Stent Thrombosis | 24 hours
  Acute stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ballabio, MD, Principal Investigator — ASST Santi Paolo e Carlo; Luca Valvassori, MD, Study Director — ASST Santi Paolo carlo
Locations (7):
- Italy (7):
  - ASST Papa Giovanni XXIII, Bergamo, Italy
  - Ospedale Bufalini, Cesena, Italy
  - Azienda Sanitaria Lecce - Ospedale "Vito Fazzi", Lecce, Italy
  - ASST Santi Paolo e Carlo, Milan, Italy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Italy
  - ASL 2 Savonese - Ospedale Santa Corona, Pietra Ligure, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Berge E, Whiteley W, Audebert H, De Marchis GM, Fonseca AC, Padiglioni C, de la Ossa NP, Strbian D, Tsivgoulis G, Turc G. European Stroke Organisation (ESO) guidelines on intravenous thrombolysis for acute ischaemic stroke. Eur Stroke J. 2021 Mar;6(1):I-LXII. doi: 10.1177/2396987321989865. Epub 2021 Feb 19. PMID 33817340
- [Background] Heck DV, Brown MD. Carotid stenting and intracranial thrombectomy for treatment of acute stroke due to tandem occlusions with aggressive antiplatelet therapy may be associated with a high incidence of intracranial hemorrhage. J Neurointerv Surg. 2015 Mar;7(3):170-5. doi: 10.1136/neurintsurg-2014-011224. Epub 2014 Nov 11. PMID 25387730
- [Background] Baek BH, Yoon W, Lee YY, Kim SK, Kim JT, Park MS. Intravenous Tirofiban Infusion After Angioplasty and Stenting in Intracranial Atherosclerotic Stenosis-Related Stroke. Stroke. 2021 May;52(5):1601-1608. doi: 10.1161/STROKEAHA.120.033551. Epub 2021 Apr 1. PMID 33793319
- [Background] Lee JI, Gliem M, Gerdes G, Turowski B, Kaschner M, Kraus B, Hartung HP, Jander S. Safety of bridging antiplatelet therapy with the gpIIb-IIIa inhibitor tirofiban after emergency stenting in stroke. PLoS One. 2017 Dec 27;12(12):e0190218. doi: 10.1371/journal.pone.0190218. eCollection 2017. PMID 29281734
- [Background] Osteraas ND, Crowley RW, Panos N, Dafer RM. Eptifibatide use following emergent carotid stenting in acute anterior circulation ischemic stroke with tandem occlusion. J Stroke Cerebrovasc Dis. 2020 Sep;29(9):105021. doi: 10.1016/j.jstrokecerebrovasdis.2020.105021. Epub 2020 Jun 17. PMID 32807436
- [Background] Delvoye F, Maier B, Escalard S, Labreuche J, Thion LA, Aknouche S, Hebert S, Redjem H, Smajda S, Ciccio G, Allard J, Sabben C, Obadia M, Maertens de Noordhout A, Olivot JM, Blanc R, Piotin M, Desilles JP, Mazighi M. Antiplatelet Therapy During Emergent Extracranial Internal Carotid Artery Stenting: Comparison of Three Intravenous Antiplatelet Perioperative Strategies. J Stroke Cerebrovasc Dis. 2021 Feb;30(2):105521. doi: 10.1016/j.jstrokecerebrovasdis.2020.105521. Epub 2020 Dec 9. PMID 33310073
- [Background] Naylor R, Rantner B, Ancetti S, de Borst GJ, De Carlo M, Halliday A, Kakkos SK, Markus HS, McCabe DJH, Sillesen H, van den Berg JC, Vega de Ceniga M, Venermo MA, Vermassen FEG, Esvs Guidelines Committee, Antoniou GA, Bastos Goncalves F, Bjorck M, Chakfe N, Coscas R, Dias NV, Dick F, Hinchliffe RJ, Kolh P, Koncar IB, Lindholt JS, Mees BME, Resch TA, Trimarchi S, Tulamo R, Twine CP, Wanhainen A, Document Reviewers, Bellmunt-Montoya S, Bulbulia R, Darling RC 3rd, Eckstein HH, Giannoukas A, Koelemay MJW, Lindstrom D, Schermerhorn M, Stone DH. Editor's Choice - European Society for Vascular Surgery (ESVS) 2023 Clinical Practice Guidelines on the Management of Atherosclerotic Carotid and Vertebral Artery Disease. Eur J Vasc Endovasc Surg. 2023 Jan;65(1):7-111. doi: 10.1016/j.ejvs.2022.04.011. Epub 2022 May 20. No abstract available. PMID 35598721
- [Background] Psychogios M, Brehm A, Lopez-Cancio E, Marco De Marchis G, Meseguer E, Katsanos AH, Kremer C, Sporns P, Zedde M, Kobayashi A, Caroff J, Bos D, Lemeret S, Lal A, Arenillas JF. European Stroke Organisation guidelines on treatment of patients with intracranial atherosclerotic disease. Eur Stroke J. 2022 Sep;7(3):III-IV. doi: 10.1177/23969873221099715. Epub 2022 Jun 3. PMID 36082254
- [Background] Turc G, Bhogal P, Fischer U, Khatri P, Lobotesis K, Mazighi M, Schellinger PD, Toni D, de Vries J, White P, Fiehler J. European Stroke Organisation (ESO) - European Society for Minimally Invasive Neurological Therapy (ESMINT) Guidelines on Mechanical Thrombectomy in Acute Ischemic Stroke. J Neurointerv Surg. 2023 Aug;15(8):e8. doi: 10.1136/neurintsurg-2018-014569. Epub 2019 Feb 26. PMID 30808653
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Turc G, Tsivgoulis G, Audebert HJ, Boogaarts H, Bhogal P, De Marchis GM, Fonseca AC, Khatri P, Mazighi M, Perez de la Ossa N, Schellinger PD, Strbian D, Toni D, White P, Whiteley W, Zini A, van Zwam W, Fiehler J. European Stroke Organisation (ESO)-European Society for Minimally Invasive Neurological Therapy (ESMINT) expedited recommendation on indication for intravenous thrombolysis before mechanical thrombectomy in patients with acute ischemic stroke and anterior circulation large vessel occlusion. J Neurointerv Surg. 2022 Mar;14(3):209. doi: 10.1136/neurintsurg-2021-018589. Epub 2022 Feb 3. PMID 35115395